CLINICAL TRIAL: NCT03184025
Title: Effect of Surface Sealant Application on Clinical Performance of HEMA Containing and HEMA-free Self-Etch Adhesives
Brief Title: Effect of Surface Sealant Application on Clinical Performance Occlusal Restorations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Neslihan Tekçe (Other)
Responsible Party: Sponsor-Investigator, Neslihan Tekçe, Faculty of Dentistry, Kocaeli University
Organization: Kocaeli University (Other)
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: 2014/239
Record Dates: First submitted 2017-06-07; First posted 2017-06-12 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Dental Caries; Class I Dental Caries; Dental Composite
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients have class I caries (Other): patients have received four restorations which included HEMA containing and HEMA-free dentin adhesive with or without surface sealing
  Interventions: Other: dentin adhesive

INTERVENTIONS:
Other: dentin adhesive — HEMA-containing and HEMA-free Self-Etch dentin adhesives clinical performance with or without surface sealant

SUMMARY:
The aim was to evaluate the clinical performance of HEMA-containing and HEMA-free all-in-one self-etch adhesives with and without a surface sealing process with a nanohybrid composite in occlusal caries restorations. The hypothesis is that the HEMA-containing and HEMA-free all-in-one self-etch adhesive and the surface sealing process would significantly effect clinical performance of occlusal restorations.

ELIGIBILITY:
Inclusion Criteria:

* patients who received four direct Class I composite restorations, those with good oral hygiene with no active periodontal or pulpal diseases, whose permanent first or second molar required restorations for occlusal carious lesions with neighboring teeth and were in occlusion with antagonist teeth, and were willing to return for follow-up examinations as outlined by the investigators.

Exclusion Criteria:

* patients with uncontrolled parafunction, those presenting with poor oral hygiene and disinterested in or refused oral hygiene instructions, molars and premolars with carious lesions on a surface other than the occlusal surface and in continuity with the occlusal cavity, pulp exposure during caries removal procedure or cavities with the risk of pulp exposure, having spontaneous pain or sensitivity to percussion, and patients with periodontal or gingival disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2014-12-29 (Actual); Study Completion 2020-12-29 (Estimated)

PRIMARY OUTCOMES:
Number of failed restorations evaluated according to the modified USPSH criteria in patients with occlusal restorations. | an average of 1 year
  In restorations, retention rate, color match, wear or loss of anatomic form, marginal discoloration, caries, marginal adaptation, and surface texture were scored success or failure according to modified United States Public Health Service (USPHS) criteria. According to this criteria, success restorations received Alfa (A) or Bravo (B) scores. Alfa (A) represents the ideal clinical situation; Bravo (B) is the clinically acceptable. Failed restorations received Charlie (C) or Delta (D) scores. Charlie (C) is the clinically unacceptable situations where the restorations had to be replaced; Delta (D) is the situation where the restoration is fractured, mobile or missing and needed to be replaced immediately.